CLINICAL TRIAL: NCT04766931
Title: A Two-part, Phase I/II, Multi-center, Double-Blind, Randomized, Vehicle-controlled Study of the Safety and Efficacy of FB2001 in Patients With Moderate to Severe Coronavirus Disease 2019 (COVID-19) Infection
Brief Title: The Safety and Efficacy of FB2001 in Healthy Subjects and Patients With COVID-19 Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Frontier Biotechnologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FB2001-102
Record Dates: First submitted 2021-02-04; First posted 2021-02-23 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Covid19
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — FB2001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- A1 FB2001 or Placebo (Experimental): single dose
  Interventions: Drug: FB2001; Drug: FB2001 Placebo
- A2 FB2001 or Placebo (Experimental): single dose
  Interventions: Drug: FB2001; Drug: FB2001 Placebo
- A3 FB2001 or Placebo (Experimental): single dose
  Interventions: Drug: FB2001; Drug: FB2001 Placebo
- A4 FB2001 or Placebo (Experimental): single dose
  Interventions: Drug: FB2001; Drug: FB2001 Placebo
- A5 FB2001 or Placebo (Experimental): single dose
  Interventions: Drug: FB2001; Drug: FB2001 Placebo
- A6 FB2001 or Placebo (Experimental): single dose
  Interventions: Drug: FB2001; Drug: FB2001 Placebo
- A7 FB2001 or Placebo (Experimental): single dose
  Interventions: Drug: FB2001; Drug: FB2001 Placebo
- B1 FB2001 or Placebo (Experimental): Once daily for 5 days
  Interventions: Drug: FB2001; Drug: FB2001 Placebo
- B2 FB2001 or Placebo (Experimental): Once daily for 5 days
  Interventions: Drug: FB2001; Drug: FB2001 Placebo
- A8 FB2001 or Placebo (Experimental): single dose
  Interventions: Drug: FB2001; Drug: FB2001 Placebo
- B3 FB2001 or Placebo (Experimental): Twice daily for 5 days
  Interventions: Drug: FB2001; Drug: FB2001 Placebo

INTERVENTIONS:
Drug: FB2001 — Subjects will be administered with FB2001 by intravenous (IV) infusion
  Other Names: DC402234
Drug: FB2001 Placebo — Subjects will be administered with FB2001 placebo by intravenous (IV) infusion
  Other Names: Placebo

SUMMARY:
This is an adaptive, Phase I/II study in 2 parts: Part 1 is to evaluate the Maximum Tolerable Dose (MTD) , tolerance, safety and pharmacokinetics of FB2001 in healthy subjects; Part 2 is to evaluate the safety, pharmacokinetics and efficacy of FB2001 in patients with moderate to severe COVID-19 disease.

DETAILED DESCRIPTION:
In Part 1 of this study, all subjects, after signing the Informed Consent Form (ICF), will be assessed during the screening phase. Only those subjects who successfully complete the screening phase and meet the study eligibility criteria will proceed to receive study treatment at the assigned doses and will be followed up for 14 days (for SAD) and 28 days (for MAD) to assess post-treatment safety.

ELIGIBILITY:
Inclusion Criteria:

Subjects are required to meet ALL of the following criteria for enrollment into the Part 1 of the study:

1. Male or female adults who are between 18 and 60 years old inclusive;
2. Weigh at least 45kg, with a BMI of 19 to 30 kg/m2 inclusive;
3. No serious underlying disease which would adversely affect the study conduct and data interpretation per the investigator;
4. Female subjects should have negative results in serum pregnancy test at screening and negative urine pregnancy test at admission:

   1. Subjects of reproductive age and their partners agree to take 2 forms of effective contraceptive measures. Note: Using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives) [e.g., hormonal contraceptives (oral, patch, injectable or vaginal ring), implantable device (implantable rod or intrauterine device), or a double barrier (e.g., diaphragm, cervical cap, oral, patch or vaginal hormonal contraceptive, condom, spermicide, or sponge)]
   2. Surgically sterile, with documentation, for at least 3 months prior to screening by one of the following means:

      Bilateral tubal ligation, Bilateral salpingectomy (with or without oophorectomy), Surgical hysterectomy, Bilateral oophorectomy (with or without hysterectomy), Postmenopausal, defined as the following: Last menstrual period greater than 12 months prior to screening
   3. Postmenopausal status confirmed by serum follicle stimulating hormone (FSH) and estradiol levels at screening
5. Agree to refrain from alcohol during the study;
6. Subjects should have normal (or abnormal but not clinically significant) laboratory results per the PI's judgement including the complete blood count, biochemistry, coagulation indices and urinalysis;
7. Subjects should have a normal (or abnormal but not clinically significant) ECG and chest X-ray at screening;
8. Subjects should be willing to cooperate and able to participate in this study, comply with all protocol requirements, and sign an informed consent;
9. Male subjects with female partners of childbearing potential must agree to use condoms for the duration of the study and until 12 weeks after completion of dosing with the study drug and must refrain from donating sperm for this same period;
10. Current non-smokers and those who have not smoked within the last 6 months. This includes the use of cigarettes, e-cigarettes, and nicotine replacement products.

Exclusion Criteria:

Subjects are required to meet NONE of the following criteria for enrollment into the Part 1 of the study:

1. HIV antibody positive;
2. HbsAg positive;
3. HCV antibody positive;
4. History of tuberculosis or lung disease as reported by subject;
5. As reported by the subject has severe cardiovascular disease, neurological disease, hematological disease, infectious disease, mental disorder, liver disease, gastrointestinal disease, lung disease, endocrine disease,immune disease or kidney disease, or has a history of the above diseases, or other symptoms known to interfere with the absorption, distribution, metabolism, or excretion of the medicine, or other conditions that the investigator believes will increase the risk of the subject and might interfere with the study conduct and results interpretation
6. Female subjects who are pregnant, lactating or have pregnancy plans in the 3 months after their study completion;
7. Subjects who participated in any other clinical study within 30 days prior to screening;
8. Subjects with known allergic reactions to the study drug or its excipients;
9. Use of any medication, including prescription or over the counter, vitamins, herbal and/or mineral supplements, dietary supplements (and/or grape fruit juice) within 14 days prior to the first treatment or during the trial, which in the opinion of the investigator may influence the trial results or the safety of the subjects:

   1. Poor venous access or issues with needle sticks, e.g., syncope
   2. Donated or lost >500 mL of blood in the previous 3 months
   3. A history of prescription drug abuse, illicit drug use within 9 months prior to screening
   4. A positive screen for alcohol or drugs of abuse at screening or admission
10. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
The Maximum Tolerable Dose (MTD) | 0~5 days
  Determination of the Maximum Tolerable Dose (MTD) of FB2001 based on the occurrence of Dose Limiting Toxicities (DLTs).
Number of participants with treatment-related adverse events as assessed by CTCAE V4.0 | 0~28 days
  Evaluation of the safety and tolerability of FB2001 after a single and multiple dose administrations in healthy volunteers.
Pharmacokinetic parameters(Cmax) | 0~5 days
  Estimate of steady state Cmax for multiple dose administration of FB2001.
Pharmacokinetic parameters(AUC0-τ) | 0~5 days
  Estimate of steady state AUC0-τ for multiple dose administration of FB2001.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Yao, Study Director — Frontier Biotechnologies Inc.
Locations (1):
- Frontage Clinical Services, Inc., Secaucus, New Jersey, United States